CLINICAL TRIAL: NCT05877079
Title: Activation of Peripheral TRPM8 Mitigates Acute Ischemic Stroke by Topically Applied Menthol
Brief Title: TRPM8 in Acute Ischemic Stroke by Topical Menthol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Collaborators: China Medical University, Taiwan (Other); Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: N202302006
Record Dates: First submitted 2023-05-14; First posted 2023-05-26 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-05

CONDITIONS: Ischemic Stroke
Keywords: TRPM8; Menthol; ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Menthol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Menthol group (Experimental): Hand and foot wraps with 8% w/w menthol lotion (20 grams each) will be delivered to each subject to wear for 5 min 5 days per week. The total duration is 4 weeks.
  Interventions: Drug: Menthol
- Non-Menthol group (Placebo Comparator): Hand and foot wraps containing the lotion (20 grams each) without menthol will be delivered to each subject to wear for 5 min 5 days per week. The total duration is 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Menthol — Patients will wear hand and foot wraps with 8% w/w menthol lotion (20 grams each) for 5 min. Patients will wear the wraps for 5 days per week. The total duration is 4 weeks.
  Arms: Menthol group
Drug: Placebo — Patients will wear hand and foot wraps with lotion without menthol (20 grams each) for 5 min. Patients will wear the wraps for 5 days per week. The total duration is 4 weeks.
  Arms: Non-Menthol group

SUMMARY:
Our previous results suggested that activation of peripheral TRPM8 expressed in the derma tissue of limbs with sufficient concentration of menthol is beneficial to stroke recovery.

In the present study, sixty patients with acute ischemic stroke were randomly divided into two groups: thirty in the treatment group and thirty in the control group. The treatment group will use an emulsion containing 8% w/w menthol, with an average of 80 grams placed inside hand and foot wraps (20 grams in each hand or foot wrap). The control group, on the other hand, will use an emulsion that does not contain any menthol, with an average of 80 grams placed inside hand and foot wraps. Participants in this study will initially undergo a detailed regular neurological examination, an assessment with the National Institutes of Health Stroke Scale (NIHSS), Barthel Index (BI) for daily living functions, and the Modified Rankin Scale (mRS) for disability. All participants will be re-evaluated after the fourth and eighth weeks of the trial, with assessments including neurological examination, NIHSS, BI, and mRS.

DETAILED DESCRIPTION:
Sixty patients with acute ischemic stroke were randomly divided into two groups: thirty in the treatment group and thirty in the control group.

Participants in this study will initially undergo a detailed regular neurological examination, an assessment with the National Institutes of Health Stroke Scale (NIHSS), Barthel Index (BI) for daily living functions, and the Modified Rankin Scale (mRS) for disability. After completing the basic assessments and signing the informed consent, participants will be randomly allocated to either the treatment group or the control group for the trial.

The treatment group will use an emulsion containing 8% w/w menthol, with an average of 80 grams placed inside hand and foot wraps (20 grams in each hand or foot wrap). Participants will wear the wraps for five minutes before removal. This process will be done once a day for five consecutive days in a week, followed by two days of rest, and will last for four weeks.

The control group, on the other hand, will use an emulsion that does not contain any menthol, with an average of 80 grams placed inside hand and foot wraps. The same procedure will be followed: participants will wear the wraps for five minutes before removal, once a day for five consecutive days in a week, followed by two days of rest, for a total of four weeks.

All participants will be re-evaluated after the fourth and eighth weeks of the trial, with assessments including neurological examination, NIHSS, BI, and mRS.

Emergency, neurology outpatient, and inpatient participants will also use the 8% w/w menthol emulsion, with an average of 80 grams placed inside hand and foot wraps (20 grams each). The same procedure will be followed: wearing the wraps for five minutes before removal, once a day for five consecutive days per week, followed by two days of rest, for a total of four weeks.

Participants will be evaluated within seven days after being diagnosed with a stroke, and then again after the fourth and eighth weeks of treatment. The evaluations will include neurological examination, NIHSS, BI, and mRS assessments.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke patients, stroke time within one week, those who are legally of age at the time of signing the consent form, NIHSS 4-20, patients who can cooperate with treatment, Self or agent agrees to sign the consent form.

Exclusion Criteria:

* NIHSS score does not meet, mRS=5, patients who cannot cooperate, moderate to severe brain trauma, pregnant women, uremia, liver cirrhosis, heart failure with pulmonary edema and coagulation dysfunction, epilepsy, alcohol, drug abuse. Participants were ranked by the investigator as unsuitable for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
NIHSS | Evaluations will be conducted within seven days of the stroke represented as the baseline data
  The National Institutes of Health Stroke Scale:a tool used by healthcare providers to objectively quantify the impairment caused by a stroke and aid planning post-acute care disposition, though was intended to assess differences in interventions in clinical trials.
NIHSS | Evaluations will be conducted at the fourth week after the start of the intervention
  The National Institutes of Health Stroke Scale:a tool used by healthcare providers to objectively quantify the impairment caused by a stroke and aid planning post-acute care disposition, though was intended to assess differences in interventions in clinical trials.
NIHSS | Evaluations will be conducted at the fourth week after the end of the intervention, i.e. the eighth week after start of intervention
  The National Institutes of Health Stroke Scale:a tool used by healthcare providers to objectively quantify the impairment caused by a stroke and aid planning post-acute care disposition, though was intended to assess differences in interventions in clinical trials.

SECONDARY OUTCOMES:
BI | Evaluations will be conducted within seven days of the stroke represented as the baseline data
  Barthel Index:It is an assessment scale used by the medical team to evaluate the patient's functional capacity in daily living. The scale is used to determine what medical care the patient needs and whether the patient is eligible for expatriate care. Lower scores on the scale indicate a patient's lack of independence.
BI | Evaluations will be conducted at the fourth week after the start of the intervention
  Barthel Index:It is an assessment scale used by the medical team to evaluate the patient's functional capacity in daily living. The scale is used to determine what medical care the patient needs and whether the patient is eligible for expatriate care. Lower scores on the scale indicate a patient's lack of independence.
BI | Evaluations will be conducted at the fourth week after the end of the intervention, i.e. the eighth week after start of intervention
  Barthel Index:It is an assessment scale used by the medical team to evaluate the patient's functional capacity in daily living. The scale is used to determine what medical care the patient needs and whether the patient is eligible for expatriate care. Lower scores on the scale indicate a patient's lack of independence.

OTHER OUTCOMES:
mRS | Evaluations will be conducted within seven days of the stroke represented as the baseline data
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
mRS | Evaluations will be conducted at the fourth week after the start of the intervention
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
mRS | Evaluations will be conducted at the fourth week after the end of the intervention, i.e. the eighth week after start of intervention
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hung Chen, PhD, Study Director — Institute of acupuncture science, College of Chinese Medicine, China Medical University
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Data including paper and electronic fileswill be destroyed after two years since the end of the study. Data obtained from the study, if digitized, will be stored on the investigator's computer in the hospital office and secured the password. Written data will be kept in a locked drawer in the investigator's office and stored separately from the subject's consent form. The data will be kept for five years after the end of the trial, at which time the digital data will be deleted from the computer and the written data will be deleted by shredder.

REFERENCES:
- [Background] Huang SS, Su HH, Chien SY, Chung HY, Luo ST, Chu YT, Wang YH, MacDonald IJ, Lee HH, Chen YH. Activation of peripheral TRPM8 mitigates ischemic stroke by topically applied menthol. J Neuroinflammation. 2022 Jul 27;19(1):192. doi: 10.1186/s12974-022-02553-4. PMID 35897101